CLINICAL TRIAL: NCT00004403
Title: Randomized Study of Albendazole in Patients With Epilepsy Due to Neurocysticercosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13286; JHUSHPH-FDR001107
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-01

CONDITIONS: Epilepsy; Cysticercosis
Keywords: cysticercosis; epilepsy; immunologic disorders and infectious disorders; neurologic and psychiatric disorders; parasitic infection; rare disease; seizures
MeSH Terms: conditions — Epilepsy; Cysticercosis; Immune System Diseases; Communicable Diseases; Neurologic Manifestations; Mental Disorders; Parasitic Diseases; Rare Diseases; Seizures | interventions — Albendazole; Dexamethasone; Phenytoin

INTERVENTIONS:
Drug: albendazole
Drug: dexamethasone
Drug: phenytoin

SUMMARY:
OBJECTIVES: I. Determine the effect of antiparasitic treatment with albendazole on the severity and duration of epilepsy due to neurocysticercosis.

II. Determine the effect of a short course of albendazole on Taenia solium cysts present in the brain.

III. Determine the natural regression of cerebral T. solium cysts in patients given placebo and their response to treatment at the end of the study.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind study. Patients are randomized to receive either albendazole and dexamethasone or placebo.

Patients receive phenytoin daily starting on day 1 and continuing until seizure free for 1 year. Albendazole and dexamethasone or placebo only is administered orally once daily on days 5-15.

Patients are asked to maintain a diary. Patients are followed on day 15 and 30, then every 3 months for 3 years.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Presence of Taenia solium infection as demonstrated by serology and head CT Head CT showing no more than 20 cysts
* At least 2 spontaneous seizures within the last 6 months excluding: Absence seizures Rolandic seizures Bilateral spike wave patterns compatible with genetic epilepsy

--Prior/Concurrent Therapy--

* No prior therapy for cysticercosis

--Patient Characteristics--

* Age: 16 to 65
* Performance status: Not specified
* Hematopoietic: Not specified
* Hepatic: Not specified
* Renal: Not specified
* Neurologic: No focal deficits No motor deficits No cranial nerve lesions History of epilepsy of less than 5 years in duration No head CT evidence of the following: Arteriovenous malformations Trauma Cerebral infarcts or hemorrhages No other focal disease not attributable to cysticercosis No moderate or severe intracranial hypertension No status epilepticus
* Other: No unstable condition due to systemic disease or cysticercosis Not pregnant

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2000-05; Study Completion 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: Robert H. Gilman, Study Chair — Johns Hopkins University